CLINICAL TRIAL: NCT03716440
Title: Using Nature Exposure Research to Reduce Impulsivity in Smokers
Brief Title: Effects of Nature Exposure on Smoking Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Lucian Conway, Professor of Social Psychology, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44-17
Record Dates: First submitted 2018-02-20; First posted 2018-10-23 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature group (Experimental): Nature exposure intervention.
  Interventions: Other: Nature exposure
- Non-nature group (Active Comparator): Non-nature exposure intervention.
  Interventions: Other: Non-nature exposure

INTERVENTIONS:
Other: Nature exposure — Participants will view images of nature.
  Arms: Nature group
Other: Non-nature exposure — Participants will view non-nature images.
  Arms: Non-nature group

SUMMARY:
Smoking continues to be the leading cause of preventable death and disease in the U.S. While smoking is a significant threat to public health in the US in general, the negative effects of smoking disproportionately affect Americans with 12 or fewer years of education and those living below the poverty line. Given these health disparities, it is vital to have widely-available treatments that can be applied in multiple contexts in a cost-efficient way. While numerous methodologies and intervention programs exist, there is a need for improved cessation programs targeted to smokers with low levels of education attainment and income, as these smokers tend to be less likely to receive cessation assistance from a health care provider or have sufficient resources to access treatments. Therefore, the present proposal aims to assess the feasibility of a tool that will improve smoking cessation programs in a short and cost-effective manner: a brief exposure to nature.

The health and wellbeing benefits of nature exposure have been well researched and are widely recognized, and research on the underlying mechanism for nature's positive impact on health has identified a reduction in impulsivity as a mediator of this effect. However, this work has never been directly translated to smoking outcomes, and thus the translational purpose of the present project is to assess the feasibility of a brief and cost-effective nature exposure intervention on smoking cessation outcomes. Prior work demonstrates the validity of the causal links in the nature -> impulsivity -> smoking cessation model. Research has shown that nature exposure reduces impulsivity for health-related outcomes, and found that increased impulsivity is linked to all stages of smoking. A necessary step in developing a practical application for this research is the aim of the present project.

Smokers will be recruited online and randomly assigned to either the Nature or Control condition. Participants in the Nature condition will be given a nature-based intervention, while participants in the Control condition will be given a non-nature-based intervention. Participants will be contacted via text message throughout the following 24 hours and asked to report their degree of urgency to smoke and number of cigarettes smoked. Participants will complete measurements of impulsivity, income, socio-economic status, and education, and additional smoking-related constructs.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least two cigarettes per day for the last seven or more days
* Must be 18 years old or older
* Must have a smart cellular phone that can send and receive text messages and open web links

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
1-item Desire to Smoke Measure | 1 day
  Self reported rating of desire to smoke. This item is scored 1 - 10 (1 = no desire to smoke; 10 = craving to smoke is extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Luke Conway, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided